CLINICAL TRIAL: NCT00339092
Title: Project Title: A RCT of HIV Adherence Case Management and Modified Directly Observed Therapy
Brief Title: Modified Directly Observed Therapy for Improving Antiretroviral Therapy Adherence in People With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Bangsberg, MD, Principal Investigator, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01MH064388 (NIH); R01MH064388 (NIH)
Record Dates: First submitted 2006-06-16; First posted 2006-06-20 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections
Keywords: HIV; ART
MeSH Terms: conditions — HIV Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Participants who receive storefront modified directly observed therapy (MDOT) of prescribed antiretrovirals
  Interventions: Behavioral: Modified Directly Observed Therapy
- Control (Active Comparator): Participants who receive standard care
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Modified Directly Observed Therapy — Treatment includes storefront modified directly observed therapy (MDOT) of prescribed antiretrovirals. Participants in the MDOT program will report to the study site each morning for 3 months, Monday through Friday, to take their HIV medication and any other medications prescribed by their primary care doctors. At the end of 3 months, participants will no longer attend the study site for medication assistance. Participants will then attend Action Point, a county program that helps participants adhere to taking medication, for an additional 3 months.
  Other Names: MDOT
  Arms: Treatment
Behavioral: Standard Care — Participants assigned to standard care will report to the study site once a month for 9 months, but will not receive any assistance with taking HIV medications. Information about medication adherence, housing, income, use of health services, drug use, sexual practices, and mental health services will be collected at each visit.
  Arms: Control

SUMMARY:
This study will evaluate the effectiveness of a modified directly observed therapy program in increasing antiretroviral therapy adherence in poor, HIV-infected residents of urban communities.

DETAILED DESCRIPTION:
Antiretroviral drug therapy (ART) is a type of medication treatment for HIV that impairs the virus's ability to multiply. When used properly, it has been shown to be successful in reducing HIV-related deaths. A 95% adherence rate to ART is required to adequately suppress the virus and prevent transmission. High rates of mental illness, substance use, and unstable housing, however, make adherence to ART particularly problematic in poor urban populations. Directly observed therapy (DOT), in which medication intake is closely monitored, improved treatment adherence during the tuberculosis epidemic of the 1990s, and is now gaining recognition as a model for improving ART adherence. HIV DOT has been successfully delivered to people residing in structured living settings. The majority of HIV-infected people, however, live outside these facilities. Therefore, there is a need for a modified version of DOT to reach HIV-infected people in community settings. This study will evaluate the effectiveness of a MDOT program in increasing ART adherence in poor, HIV-infected residents of urban communities.

Participants in this open label study will be randomly assigned to either receive standard care or participate in the MDOT program. Participants assigned to standard care will report to the study site once a month for 9 months, but will not receive any assistance with taking HIV medications. Information about medication adherence, housing, income, use of health services, drug use, sexual practices, and mental health services will be collected at each visit. Participants in the MDOT program will report to the study site each morning for 3 months, Monday through Friday, to take their HIV medication and any other medications prescribed by their primary care doctors. If an individual does not attend a visit, study staff will try to locate the individual in the neighborhood to deliver the medication. Medication for the weekend will be prepared by study staff, but participants will take it on their own at home. At the end of 3 months, participants will no longer attend the study site for medication assistance. They will, however, participate in Action Point, a county program that helps participants adhere to taking medication, for an additional 3 months. Participants will also check in with the study staff once a month. Following this, participants may choose to discontinue the Action Point program for the final 3 months of the study. They will continue monthly check-in visits with the study staff. At each visit, interviews will be conducted and medication adherence will be assessed. Blood tests will be performed once every 3 months throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Severely immunosuppressed (HIV viral load of greater than 400 copies/ml)
* Does not consistently take prescribed ARV
* Currently prescribed HIV medications or prescribed to start taking HIV medications

Exclusion Criteria:

* Currently participating in any other adherence program or intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
CD4 and Viral Load | Measured at baseline and Months 3, 6, and 9

SECONDARY OUTCOMES:
Adherence | Measured monthly for 9 months

CONTACTS AND LOCATIONS:
Overall Officials: David R. Bangsberg, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- UCSF Market Street Study Site, San Francisco, California, United States